CLINICAL TRIAL: NCT06863961
Title: A Phase II, Multicenter, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of RO7790121 in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of Afimkibart (RO7790121) in Participants With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS45570; 2024-515494-95-00 (Other: EU CT Number)
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Afimkibart Group I (Experimental): Participants will receive afimkibart via subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Afimkibart Group II (Experimental): Participants will receive afimkibart via SC injection.
  Interventions: Drug: Afimkibart
- Afimkibart Group III (Experimental): Participants will receive afimkibart via SC injection.
  Interventions: Drug: Afimkibart
- Placebo (Placebo Comparator): Participants will receive placebo via SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as SC injection.
  Other Names: PF-06480605; RVT-3101; RO7790121
  Arms: Afimkibart Group I; Afimkibart Group II; Afimkibart Group III
Drug: Placebo — Placebo will be administered as SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Afimkibart (also known as RO7790121) in participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* AD diagnosis confirmed by a dermatologist according to the Hanifin/Rajka criteria at least 1 year prior to screening
* Moderate to severe AD
* At least once daily use of an additive-free, bland emollient for at least 7 days prior to the baseline visit and during the study

Exclusion Criteria:

* Evidence of other skin conditions that would interfere with the assessment of AD, including, but not limited to, for example cutaneous T-cell lymphoma, allergic contact dermatitis
* IV, IM, IL, and oral corticosteroids (inhaled, ophthalmic drops, and nasal corticosteroids are allowed) within 4 weeks of the baseline visit and during the study
* Topical treatment for AD including, but not limited to topical corticosteroids, topical calcineurin Inhibitors, topical PDE-4 inhibitors, , prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea or filaggrin within 7 days prior to the baseline visit and during the study
* Any active infection or other active skin diseases that required treatment with parenteral anti-infectives within 4 weeks or oral anti-infective treatment within 2 weeks prior to baseline
* Acquired or congenital immunodeficiency
* Systemic therapies that are also used in the treatment of AD, including, but not limited to methotrexate, cyclosporine, azathioprine, mycophenolate mofetil within 4 weeks of the baseline visit and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Eczema Area and Severity Index-75 (EASI-75) Response (>= 75% Improvement from Baseline) at Week 16 | Baseline and Week 16

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Investigator Global Assessment (IGA) Score of Clear (0) or Almost Clear (1) with >= 2-Grade Improvement at Week 16 and Week 32 | At Week 16 and Week 32
Percentage of Participants who Achieve EASI-75 Response at Week 32 | At Week 32
Percentage of Participants who Achieve EASI-90 Response at Week 16 and Week 32 | At Week 16 and Week 32
Percent Change from Baseline in EASI by Visit | Baseline up to end of study (approximately 1 year)
Percent Change from Baseline in Peak Pruritus Numerical Rating Scale (NRS) Score by Visit | Baseline up to end of study (approximately 1 year)
Change from Baseline in Dermatology Quality of Life Index at Week 16, Week 32 and by Visit | Baseline, weeks 4, 10, 16, 22 and 32
Percentage of EASI-75 Responders at Week 16 | At Week 16
Percentage of Participants with Adverse Events | Baseline up to end of study (approximately 1 year)
Serum Concentration of Afimkibart at Specified Timepoints | Weeks 0, 2, 4, 6, 10, 14, 16, 18, 22, 26, 30, 32 and monthly at weeks 4, 8 and 12 after treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- United States (21):
  - University of California Los Angeles, Los Angeles, California
  - Dermatology Research Associate, Los Angeles, California
  - Suncoast Research Associates LLC - ERN - PPDS, Doral, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Dermatology Affiliates Research Institute, LLC, Atlanta, Georgia
  - Dawes Fretzin Clinical Res LLC, Indianapolis, Indiana
  - Revival Research Institute, LLC, Troy, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Care Access Research - Hoboken, Hoboken, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Centricity Research Dublin, Dublin, Ohio
  - DOCS Clinical Research - Springfield, Springfield, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Best Skin Research LLC, Camp Hill, Pennsylvania
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Cumberland Skin Center for Clinical Research LLC, Hermitage, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Modern Research Associates, Dallas, Texas
  - Reveal Research Institute, Dallas, Texas
  - Care Access Research - Arlington, Arlington, Virginia
- Brazil (6):
  - Centro de Pesquisas da Clínica IBIS, Salvador, Estado de Bahia
  - Centro de Estudos em Terapias Inovadoras ? CETI, Curitiba, Paraná
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Centro de Pesquisa São Lucas, Campinas, São Paulo
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A, Rio de Janeiro
- Canada (8):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Centricity Research, London, Ontario
  - DermEffects, London, Ontario
  - Lynde Institute for Dermatology, Markham, Ontario
  - DermEdge, Mississauga, Ontario
  - Ryan Clinical Research Inc, Newmarket, Ontario
  - Centre de Recherche Saint-Louis, Québec
- France (2):
  - Hopital Charles Nicolle, Rouen, Nord
  - Hopital Saint Louis, Cedex 10, Paris
- Germany (6):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinisches Studienzentrum, Bad Bentheim, Lower Saxony
  - DRK Krankenhaus Chemnitz-Rabenstein, Chemnitz, Saxony
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg, Saxony-Anhalt
  - CRS Clinical Research Services Kiel GmbH, Kiel, Schleswig-Holstein
  - Dermatologikum Hamburg GmbH, Hamburg
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Emilia-Romagna
  - Fondazione IRCCS CA? Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico Gaspare Rodolico - San Marco (Presidio G. Rodolico), Catania, Sicily
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
- Poland (12):
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Pratia Katowice I, Katowice
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow
  - Specjalistyczny Gabinet Dermatologiczny dr n. med. Pawel Brzewski, Krakw
  - Dermoklinika, Lodz
  - Uniwersytecki Szpital Kliniczny im.Fryderyka Chopina w Rzeszowie, Rzeszów
  - LASER CLINIC S.C. Dr Tomasz Kochanowski Dr Andrzej Krolicki, Szczecin
  - MICS Centrum Medyczne Torun, Torun
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago., Santiago de Compostela, LA Coruna
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing